CLINICAL TRIAL: NCT01046578
Title: Aromatase Inhibitor Effects on Ovarian Function During the Follicular and Early Luteal Phase in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Roger Pierson, PhD, University of Saskatchewan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WHIRL-08-1200
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Fertility
Keywords: Folliculogenesis; Letrozole; Aromatase Inhibitor; Estrogen
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Single Dose 12mm follicle (Experimental): Single dose (20mg) of an aromatase inhibitor (Letrozole/Femara(TM); n = 10) initiated at follicle diameter of 12 mm
  Interventions: Drug: Letrozole
- Single Dose 18mm follicle (Experimental): Single dose (20mg) of an aromatase inhibitor (Letrozole/Femara(TM); n = 10) initiated at follicle diameter of 18 mm
  Interventions: Drug: Letrozole
- Single Dose Post Ovulation (Experimental): Single dose (20mg) of an aromatase inhibitor (Letrozole/Femara(TM); n = 10) initiated 24-48 post ovulation
  Interventions: Drug: Letrozole
- Multi Dose 12mm follicle (Experimental): Multi dose (2.5mg/day for 5 days) of an aromatase inhibitor (Letrozole/Femara(TM); n = 10) initiated at follicle diameter of 12 mm
  Interventions: Drug: Letrozole
- Multi Dose 18mm follicle (Experimental): Multi dose (2.5mg/day for 5 days) of an aromatase inhibitor (Letrozole/Femara(TM); n = 10) initiated at follicle diameter of 18 mm
  Interventions: Drug: Letrozole
- Multi Dose Post Ovulation (Experimental): Multi dose (2.5mg/day for 5 days) of an aromatase inhibitor (Letrozole/Femara(TM); n = 10) initiated 24-48 hours post ovulation
  Interventions: Drug: Letrozole
- Control (No Intervention): No intervention given, followed for course of study on a natural cycle

INTERVENTIONS:
Drug: Letrozole — 20 mg, one tablet a day for one day, starting on the day the dominant follicle reaches 12 mm in diameter
  Other Names: Femara (TM)
  Arms: Single Dose 12mm follicle
Drug: Letrozole — 20 mg, one tablet a day for one day, starting on the day the dominant follicle reaches 18 mm in diameter
  Other Names: Femara (TM)
  Arms: Single Dose 18mm follicle
Drug: Letrozole — 20 mg, one tablet a day for one day, starting 24-48 hours after ovulation of the dominant follicle is observed
  Other Names: Femara (TM)
  Arms: Single Dose Post Ovulation
Drug: Letrozole — 2.5 mg, one tablet a day for five days, starting 24-48 hours after ovulation of the dominant follicle is observed
  Other Names: Femara (TM)
  Arms: Multi Dose Post Ovulation
Drug: Letrozole — 2.5 mg, one tablet a day for five days, starting on the day the dominant follicle reaches 18 mm in diameter
  Other Names: Femara (TM)
  Arms: Multi Dose 18mm follicle
Drug: Letrozole — 2.5 mg, one tablet a day for five days, starting on the day the dominant follicle reaches 18 mm in diameter
  Other Names: Femara (TM)
  Arms: Multi Dose 12mm follicle

SUMMARY:
A single center, open label randomized clinical trial designed to examine ovarian follicular dynamics following attempted atresia induction during the late follicular and early luteal phase of the menstrual cycle using an aromatase inhibitor.

We hypothesize that administration of an aromatase inhibitor (AI) at biologically important times of the natural menstrual cycle will cause ovulatory failure in women with preovulatory follicles and failure of luteogenesis in women who have recently ovulated. It is proposed that atresia of the dominant follicle and formation of anovulatory structures will be associated with arrested endometrial development and a shortened interval to menstrual bleeding (3 days). We anticipate that this will provide us with information to facilitate the development of a new method for emergency contraception and a greater understanding of human folliculogenesis.

The rationale for the proposed research project is based on the ovarian synchronization concepts developed and documented in the bovine model in the Reproductive Science and Medicine Research group at the University of Saskatchewan combined with novel human ovarian wave concepts of folliculogenesis first elucidated in the Women's Health Imaging Research Laboratory (WHIRL) in the Department of Obstetrics, Gynecology and Reproductive Sciences.

DETAILED DESCRIPTION:
In clinical practice emergency contraception (EC) intends to suppress follicular development, ovulation, or the ability of a conceptus to implant. Exogenous steroids, estrogen and progestin, are used in various formulations to accomplish the suppression. Though EC are now available 'over-the-counter' in Canada and many countries around the world; the ovarian response is unpredictable and EC do not inhibit ovulation at the most critical times of the menstrual cycle. In 2002 approximately 120,000 of 450,000 pregnancies in Canada ended in elective pregnancy termination. In the US 49% of the 3.5 million annual pregnancies were unintended and 54% of the unintended pregnancies resulted in elective termination.

Current hormonal contraceptive regimens, pre and post coital, are based on the traditional theory of follicular development that states that a single group of antral follicles is recruited in the late luteal phase for growth. Recent documentation has show that human ovarian folliculogenesis occurs in a 2-3 wave like pattern during a menstrual cycle. Wave emergence has been documented to occur in the early luteal phase with the final wave being ovulatory. The new model of follicular wave dynamics is well established and supported by experimental evidence in the bovine and equine models.

Traditionally these hormonal medications are taken 72 to 120 hours after known or suspected barrier contraception failure or unprotected intercourse. The two standard steroidal EC methods are Plan BTM, containing of 0.75 mg levonorgestrel (LNG), and the Yuzpe method, containing 0.1 mg ethinyl estradiol (EE) and 0.5 mg LNG. Ovarian follicular development and ovulation in women have been studied after EC use; however, the mechanisms underlying follicular growth, regression, and ovulation during EC use remain poorly elucidated. The mechanism of action differs with each EC regimen as well as being dependent upon the relative timing between dosing, intercourse, and ovulation. Previous studies have shown that EC are most effective if used when the dominant follicle diameter is small (4 to 5 days prior to ovulation), however, during this time interval intercourse is less likely to result in pregnancy whether or not EC were administered.

All current emergency contraception (EC) options are guided by the traditional theory of follicular development. Based on the findings of an unpredictable response of the ovaries to EC treatment, the occurrence of ovulation after treatment with EC, and findings of follicle growth in a 2-3 wave pattern, we need to reconsider the phase of the menstrual cycle and the treatment given for emergency contraception.

Aromatase inhibitors (AI) prevent the enzymatic conversion of androgens to estrogens. This significantly lowers serum estrogen levels. AI have been administered around the time of menses for ovulation induction and ovulation was seen to follow 10 to 12 days later. The rationale for inducing atresia of dominant follicles stems from this observation. Acute estradiol deprivation should theoretically initiate atresia of all viable follicles in the cohort resulting in the emergence of a new follicle wave without an ovulation event occurring.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential with normal reproductive function;
* Women between 18 and 35 years of age;
* Normal Body Mass Index (18-30);
* Are naïve to OC or have discontinued OC at least 2 months prior to study entry;
* Subject has signed the informed consent form;
* Subject is in good general health as confirmed by medical history and physical examination

Exclusion Criteria:

* Irregular menstrual cycles;
* Any contraindication for oral contraception use;
* Known hypersensitivity to Letrozole and co-administered medications;
* Evidence of Polycystic Ovary Syndrome (PCOS) or Endometriosis;
* History of pituitary tumor;
* Pregnancy (suspected or diagnosed) or lactation;
* HIV, HBV, HCV infection;
* Vaginal infection;
* Abnormal ECG;
* Abnormal lab tests for blood profile, liver function and renal function;
* Uncontrolled diabetes and blood pressure;
* History or suspicion of alcohol or drug abuse;
* History of severe mental disorders;
* Participation in an investigational drug trial in the 30 days prior to selection;
* A subject who exhibits a disorder that is a contraindication to steroid hormonal therapy, including, for example, the following conditions:
* History of/or actual thrombophlebitis or thromboembolic disorders.
* History of/or actual cerebrovascular disorders.
* History of/or actual myocardial infarction or coronary arterial disease.
* Active liver disease or history of/or actual benign or malignant liver tumors.
* Known or suspected carcinoma of the breast.
* Known or suspected oestrogen-dependent neoplasia.
* Undiagnosed abnormal vaginal bleeding
* Any ocular lesion arising from ophthalmic vascular disease, such as partial or complete loss of vision or defect in visual fields.
* Smokes.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
fate of the dominant follicle or luteal structure | 40-45 days

SECONDARY OUTCOMES:
interval to follicle wave emergence, and interval to selection of a dominant follicle | 40-45 days
endometrial thickness/pattern | 40-45 days
ultrasonographic image attributes of follicular structures that develop after administration of treatment | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Pierson, PhD, Principal Investigator — University of Saskatchewan; Donna R Chizen, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Allaway HC, Chizen DR, Adams GP, Pierson RA. Effects of a single 20 mg dose of letrozole on ovarian function post dominant follicle selection: an exploratory randomized controlled trial. J Ovarian Res. 2017 Jan 21;10(1):6. doi: 10.1186/s13048-017-0303-x. PMID 28107821